CLINICAL TRIAL: NCT03586323
Title: Awake Fiber Optic Intubation (AFOI) in Patients With Stenosis of the Upper Airway: Utility of the Laryngeal Nervous Block
Brief Title: Awake Fiber Optic Intubation (AFOI) and Laryngeal Nervous Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Alessandri, Principal Investigator, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AFOISUA
Record Dates: First submitted 2018-06-29; First posted 2018-07-13 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Airway Complication of Anesthesia
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-SLNB (Experimental): performed a superior laryngeal nerve block with lidocaine
  Interventions: Drug: superior laryngeal nerve block with lidocaine
- S-SLNB (Placebo Comparator): performed a superior laryngeal nerve block with saline
  Interventions: Drug: superior laryngeal nerve block with lidocaine

INTERVENTIONS:
Drug: superior laryngeal nerve block with lidocaine — SLNB was performed with 4 ml of 1.5% lidocaine below the thyroid membrane
  Other Names: L-SLNB

SUMMARY:
Oncologic laryngeal surgery is a challenge for anesthesiologists and awake fiberoptic intubation (AFOI) is mandatory to manage difficult airways and prevent the Can't Intubate Can't Oxigenate (CICO). Laryngospasm and oversedation are dangerous complication often life-threatening in this kind of patient. Superior laryngeal nerve block (SLNB) could be an alternative technique useful to reduce risks and to improve patient comfort. Aim of this study is to assess the procedural comfort of the SLNB during AFOI, in a population of patients suffering from severe airways obstruction undergoing pharyngeal-laryngeal surgery. 40 patients will be randomized in two groups(20 for each group) and will be treated with continuous infusion of remifentanil, topic anesthesia of the base of the tongue and intercricoid block. In group A will be associated the SLNB; placebo will be administered in group B.

DETAILED DESCRIPTION:
Patients will be randomized in two groups: group A: treated with continuous infusion of remifentanil, topic anesthesia of the base of the tongue, intercricoid block and SLNB; group B: treated with continuous infusion of remifentanil, topic anesthesia of the base of the tongue and intercricoid block. After the first measurement of vital parameters (T0), patients will received a continuous intravenous infusion of remifentanil at a rate ranged between 0.05 and 0.15 mcg/kg/min, reached by titration of a conscious sedation plane corresponding to the 0/-1 stage of the RASS scale. In all patients of both groups topical anesthesia of the oropharynx mucosa will be performed through 10 puffs of 10% lidocaine spray at the back of the tongue and at the base of the palatopharyngeal and palatoglossal arch. In Group A SLNB will be performed by administering 4 ml of 1.5% lidocaine below the thyroid membrane, which is palpated in addition to the intercricoid block by translaringeal puncture and 4 ml of lidocaine 1,5%. In group B intercricoid block will be performed by translaringeal puncture and 4 ml of 1.5% lidocaine. Group B will receive placebo instead of the regional block. After regional anesthesia, the patient will be placed on the operating table with the head in a neutral position. The vital parameters and the level of sedation reached (T1) will be registered. If SpO2 will be less than 96%, the patient will be pre-oxygenated with FiO2 100%. AFOI procedure will be performed using a 4 mm Olympus LF-2 bronchoscope and spiral tracheal tubes (internal diameter of between 5-6 mm) will be used. Discomfort during AFOI will be evaluated through the Fiber Optic Intubation Comfort Score. During AFOI procedure, unstructured airway maneuvers (neck's hyperextension, jaw subluxation, and pulling the tongue manually) will be evaluated. Hypoxemia, aspiration of secretions and time to perform intubation will be reported.

After intubation, a new evaluation of the vital parameters will be performed (T2) and patients will undergo to a total intravenous general anesthesia in accordance with the current international protocols. The primary endpoint will be to evaluate if SLNB is able to reduce the degree of discomfort of the AFOI procedure measured with the relative risk of Fiber Optic Intubation Comfort Score > 1. Secondary endpoint will be incidence of hypoxemia, time required to intubate, intraprocedural hemodynamic stability, airway obstruction score, need to aspirate secretions during AFOI, Tracheal Tube Tolerance Score.

ELIGIBILITY:
Inclusion Criteria:

* aged >18 years
* undergoing elective AFOI for upper airway obstruction

Exclusion Criteria:

* patients with respiratory tirage and cornage
* Arnè multifactorial scale < 11

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-15 (Actual); Primary Completion 2018-07-24 (Estimated); Study Completion 2018-08-01 (Estimated)

PRIMARY OUTCOMES:
discomfort | up to 10 minutes
  to evaluate if SLNB is able to reduce the degree of discomfort of the AFOI procedure measured with the relative risk of Fiber Optic Intubation Comfort Score > 1

SECONDARY OUTCOMES:
incidence of hypoxemia | up to 10 minutes
  number of desaturation events
time required to intubate | up to 10 minutes
  minutes to intubation
intraprocedural hemodynamic stability | up to 10 minutes
  reducing blood pressure > 30%

CONTACTS AND LOCATIONS:
Locations (1):
- Sapienza University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No